CLINICAL TRIAL: NCT00614289
Title: Phase 1 Study to Demonstrate Efficacy of Epikeia Coatings in a Human Clinical Trial
Brief Title: Novel Topical Treatment of Hand Dermatitis (Eczema)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Adelaide A. Hebert, MD, University of Texas Health Science Center-Houston, Dermatology Clincial Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-06-0347; NIH Grant 1R43AR525441-1A1
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2008-10

CONDITIONS: Contact Dermatitis; Eczema, Contact
Keywords: Mild to Moderate Hand Dermatitis; Hand Eczema
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Epikeia Coatings — Topical skin coating

SUMMARY:
This study is designed as a prospective, randomized, double-blind right/left comparison of Epikeia coatings to improve hand dermatitis.

DETAILED DESCRIPTION:
Hand dermatitis was chosen for investigation due to high incidence and typical symmetrical involvement that allows for right/left treatment comparisons. Hand dermatitis is also important due to its implication on healthcare workers in particular, where frequent hand washing and chronic occlusion from gloving, provide a route for skin sensitization to natural rubber latex proteins increase the risk of colonization of microorganisms on the skin, and thereby increase the likelihood of contact dermatitis.

This feasibility study will be performed to evaluate the efficacy of PVDF coatings in treating chronic hand dermatitis.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following inclusion criteria:

1. 18 years of age or older;
2. have mild to moderate hand dermatitis, according to Investigator Global Assessment (see below);
3. be generally healthy, as determined by brief medical history;
4. have a negative urine test for pregnancy if female, and use of highly effective method of birth control, such as condoms & spermacide, implants, injectables, combined oral contraceptives, intrauterine device (IUD's), sexual abstinence, or a vasectomized partner. For subjects using a hormonal contraceptive method, [i.e., birth control pill (BCP)], the dose and type of BCP should stay constant 1 month prior to enrollment and throughout the study, and
5. be capable of understanding and signing the consent form.

Exclusion Criteria:

Subjects will be excluded from the study if they:

1. have clinically relevant allergic or irritant contact dermatitis and the inability to avoid exposure;
2. have severe and very severe hand dermatitis according to the Investigator Global Assessment;
3. have severe vesiculation or bullae;
4. have a history of psoriasis, contact urticaria, and/or pustular diseases of the hands;
5. have had therapy of the hands with potent topical corticosteroids within one month of enrollment;
6. have used systemic treatment with oral retinoids, corticosteroids, or with PUVA within the 8 week period prior to the beginning of the study
7. have a history of alcoholism or drug abuse;
8. have a history or current evidence of a chronic or infectious skin disease; and
9. are pregnant or lactating females, or using method of birth control that does not comply with highly effective methods of birth control listed under inclusion criteria; Pregnant or lactating females, or using method of birth control that does not comply with highly effective methods of birth control listed under inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The endpoints for evaluation will be the within subject (test vs. control hands) comparison on Investigator Global Assessment, and Hand Eczema Area and Severity Scores. | 85 Days

SECONDARY OUTCOMES:
Ordinal scales measuring subjective efficacy, pain and itching. | 85 Days

CONTACTS AND LOCATIONS:
Overall Officials: Adelaide A. Hebert, MD, Principal Investigator — University of Texas Health Science Center, Department of Dermatoloy
Locations (1):
- UTHSC Houston, Dermatology Clincial Research Center, Houston, Texas, United States